CLINICAL TRIAL: NCT06414629
Title: Implementation and Evaluation of Simulation-Based Mentorship Program (SBMP) in Nepal Using the RE-AIM Framework
Brief Title: An Implementation Research of Simulation Based Mentorship Program
Acronym: SBMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: One Heart Worldwide (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OHW1
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Maternal Health; Neonatal Health
Keywords: Simulation; Mentorship; Capacity building

STUDY DESIGN:
Intervention Model Description: The study Birthing Centers were categorized into Intervention Birthing Center and Control Birthing Center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group/ Intervention Birthing Center (Experimental): The nurses working in the Intervention Birthing Centers received the Simulation Based Mentorship Program.
  Interventions: Other: Simulation Based Mentorship Program
- Control Group/ Control Birthing Center (No Intervention): The nurses working in the Intervention Birthing Centers did not receive the Simulation Based Mentorship Program.

INTERVENTIONS:
Other: Simulation Based Mentorship Program — In this program, local level mentors were developed to provide regular mentorship on low-dose high-frequency approach in contrast to one-time coaching in a long gap. This program combined the existing package of the continuum of care along with Helping Babies Survive (HBS) & Helping Mothers Survive (HMS) guidelines, adopting a simulation-based onsite mentoring and coaching approach. The mentors provided monthly mentorship on following seven modules topics to the nurses of the intervention birthing centers:
  1. Infection prevention
  2. Antenatal care and counseling
  3. Essential care of labor and birth
  4. Helping babies breathe
  5. Bleeding after birth
  6. Essential care of labor and birth
  7. Postnatal care and counseling
  Every monthly session was followed by four weekly practice sessions. The nurses from intervention birthing centers were also called mentees.
  Other Names: SBMP
  Arms: Intervention Group/ Intervention Birthing Center

SUMMARY:
The goal of this research was to evaluate the effectiveness and implementation outcomes of the Simulation Based Mentorship Program (SBMP) which was implemented in four districts of Nepal. The main questions it aims to answer are:

1. What is the reach of the Simulation Based Mentorship Program?
2. What is the effect of Simulation Based Based Mentorship Program on knowledge, clinical skills, and confidence of nurses working in Birthing Centers of four district of Nepal?
3. How was the program adopted by the Birthing Centers?
4. How was the program implemented?
5. What is the perception regarding the maintenance of the program?

The nurses working in the Birthing Centers were the study participants, and they received simulation-based monthly mentorship on following seven modules related to essential obstetric and newborn care every month:

1. Infection prevention
2. Antenatal care and counseling
3. Essential care of labor and birth
4. Helping babies breathe
5. Bleeding after birth
6. Pre-eclampsia and eclampsia management
7. Postnatal care and counseling

DETAILED DESCRIPTION:
As the evidence showed gaps in the knowledge and skills of existing maternal and newborn health providers, we designed a Simulation-Based Mentorship Program (SBMP) to bridge the gaps. In this program, local-level mentors were developed to provide regular mentorship using a low-dose high-frequency approach in contrast to one-time coaching in a long gap. This program combined the existing package of the continuum of care along with Helping Babies Survive (HBS) & Helping Mothers Survive (HMS) guidelines, adopting a simulation-based onsite mentoring and coaching approach.

The main aim of this mentorship program was to improve the quality of essential obstetric and newborn care provided by the nurses and Auxiliary Nurse Midwives (ANMs) irrespective of their pre-service and in-service training exposure by identifying gaps, providing regular technical support on the site, building close relationships between mentors and mentees, and increasing communication, backed up by regular practice in simulation labs to help in skill retention. In this mentorship program, mentorship was provided to both the Skilled Birth Assistants (SBAs) and non-Skilled Birth Attendants in their workstations to capacitate them in promoting mother and newborn health outcomes.

Reach, Effectiveness, Adoption, Implementation, and Maintenance (REAIM) Dimensions in the study were:

Reach

1. Number and percentage of Birthing centers intervened in the district
2. Number and percentage of nurses trained as district-level mentors
3. Number and percentage of nurses (and Auxiliary Nurse Midwives) receiving the intervention (simulation-based mentorship)
4. Perception regarding the representativeness of participants in the program

Effectiveness

1. Immediate change in knowledge, skills, and confidence (midline results)- compared with control group
2. Perceived reasons for program effectiveness

Adoption

1. Number and percentage of intervention sites completing all 6 monthly sessions
2. Number and percentage of mentees participating in all 6 monthly sessions
3. Number and percentage of mentees participating in weekly sessions
4. Reasons for participation/ non-participation

Implementation

1. Plan vs. actual implementation (duration between monthly sessions)
2. Perception regarding various components of the program (content, teaching and learning methods, mentors)
3. Challenges encountered during implementation, adaptations made/ mitigation measures adopted

Maintenance

1. Number and percentage of mentors and mentees remaining after 4 to 6 months of Simulation Based Mentorship Program (SBMP) implementation (end-line)
2. Retention of knowledge, skills, and confidence 4 to 6 months after completion of the intervention (end-line results) compared with the control group
3. Capital cost and recurrent cost required for continuation at government level
4. Application of learnings in a real setting (during and after the program implementation)
5. Willingness to implement the program in the health facilities of Simulation Based Mentorship Program (SBMP) implemented local levels after completion of the intervention
6. Continuation of mentoring/ learning in the simulation labs/ using manikins after completion of monthly sessions by mentors and mentees
7. Challenges and recommendations for continuation

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in selected Birthing Centers during the baseline enrollment

Exclusion Criteria:

* Newly recruited nurses by the Birthing Centers

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge, confidence and skills on seven modules | 1 year
  The knowledge and confidence scores of intervention and control group's nurses in all seven modules were compared before and after the study. However, skills scores of seven modules were measured only in intervention group's nurses. The overall maximum obtainable score was 127 points for knowledge assessment, 210 points for confidence assessment, and 340 points for skills assessment. The scores obtained by the participants were expressed as percentage, and a mean score was calculated for each module. A score of 80% or more was considered to be appropriate. High scores indicated better outcome, and low scores indicated poor outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Surya Bhatta, MHCDS, Study Director — One Heart Worldwide
Locations (1):
- One Heart Worldwide, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Utz B, Siddiqui G, Adegoke A, van den Broek N. Definitions and roles of a skilled birth attendant: a mapping exercise from four South-Asian countries. Acta Obstet Gynecol Scand. 2013 Sep;92(9):1063-9. doi: 10.1111/aogs.12166. Epub 2013 Jun 15. PMID 23656549
- [Background] Olson KR, Caldwell A, Sihombing M, Guarino AJ, Nelson BD, Petersen R. Assessing self-efficacy of frontline providers to perform newborn resuscitation in a low-resource setting. Resuscitation. 2015 Apr;89:58-63. doi: 10.1016/j.resuscitation.2015.01.008. Epub 2015 Jan 19. PMID 25613363
- [Background] Alamrani MH, Alammar KA, Alqahtani SS, Salem OA. Comparing the Effects of Simulation-Based and Traditional Teaching Methods on the Critical Thinking Abilities and Self-Confidence of Nursing Students. J Nurs Res. 2018 Jun;26(3):152-157. doi: 10.1097/jnr.0000000000000231. PMID 29016466
- [Background] Krielen P, Meeuwsen M, Tan ECTH, Schieving JH, Ruijs AJEM, Scherpbier ND. Interprofessional simulation of acute care for nursing and medical students: interprofessional competencies and transfer to the workplace. BMC Med Educ. 2023 Feb 11;23(1):105. doi: 10.1186/s12909-023-04053-2. PMID 36774481
- [Background] Barre J, Michelet D, Truchot J, Cabon P, Tesniere A. Midwifery students' retention of learning after screen-based simulation training on neonatal resuscitation: a pilot study. BMJ Simul Technol Enhanc Learn. 2020 Apr 6;7(1):31-34. doi: 10.1136/bmjstel-2019-000525. eCollection 2021. PMID 35521074
- [Background] Cant RP, Cooper SJ. Use of simulation-based learning in undergraduate nurse education: An umbrella systematic review. Nurse Educ Today. 2017 Feb;49:63-71. doi: 10.1016/j.nedt.2016.11.015. Epub 2016 Nov 22. PMID 27902949
- [Background] Lee BO, Liang HF, Chu TP, Hung CC. Effects of simulation-based learning on nursing student competences and clinical performance. Nurse Educ Pract. 2019 Nov;41:102646. doi: 10.1016/j.nepr.2019.102646. Epub 2019 Oct 23. PMID 31698255
- [Background] Hung CC, Kao HS, Liu HC, Liang HF, Chu TP, Lee BO. Effects of simulation-based learning on nursing students' perceived competence, self-efficacy, and learning satisfaction: A repeat measurement method. Nurse Educ Today. 2021 Feb;97:104725. doi: 10.1016/j.nedt.2020.104725. Epub 2020 Dec 16. PMID 33373813